CLINICAL TRIAL: NCT00635206
Title: Investigation of a Novel Positive Pressure Therapy to Rescue Patients Failing to Tolerate CPAP During an Initial Encounter
Acronym: BIPAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clayton Sleep Insititute (Industry)
Responsible Party: Eric Powell, PH. D, Clayton Sleep Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIPAP Rescue; ABF-2007-MCT-03
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Auto M series device set to Bi Flex
  Interventions: Device: BiPap auto with Fi Flex
- 2 (Active Comparator): Set to standard CPAP
  Interventions: Device: Standard CPAP

INTERVENTIONS:
Device: BiPap auto with Fi Flex — * MinEPAP = 4 cmH2O for prescribed CPAP ≤ 10 cmH2O (use 6 cmH2O for prescribed CPAP > 10 cmH2O)
  * MaxIPAP = 25 cm H2O
  * MinPS = 2 cm H2O (cannot be adjusted)
  * MaxPS = 8 cm H2O
  * Bi-Flex setting of 3
  Arms: 1
Device: Standard CPAP — CPAP ≤ 10 cmH2O (use 6 cmH2O for prescribed CPAP > 10 cmH2O)
  Arms: 2

SUMMARY:
The primary objective outcome is the proportion of participants compliant (at least four hours of use per night for all nights) in the Auto Bilevel group compared to the CPAP group after 90 days of treatment during the investigation. Proportion will be calculated using the cumulative number of hours on therapy divided by the total number of days of the investigation for each participant. The mean and standard deviation of these mean therapy hours will then be calculated for each arm of the investigation. Participants with compliance of at least four hours will be classified as "compliant" and those with less than four hours will be classified as "non-compliant". The null hypothesis will be rejected if the mean of the primary objective outcome for all participants in the BiPAP® Auto with Bi-Flex® therapy arm is significantly greater than that for all participants in the CPAP therapy arm.

Secondary Measures

The secondary measures used to evaluate potentially improved adherence to BiPAP® Auto with Bi-Flex® therapy compared to CPAP therapy will include:

* Hours of use per night, for all nights
* Hours of use per night, for nights with therapy use
* Device derived AHI
* Heart Rate Variability
* Functional Outcomes of Sleep Questionnaire (FOSQ),
* 10 cm Visual Analog Scale (VAS) for mask comfort and satisfaction with therapy,
* Epworth Sleepiness Scale (ESS) questionnaire
* Psychomotor Vigilance Task
* Attitudes toward use
* Actigraphy (sleep continuity) and sleep diary
* Fatigue Severity Scale
* Daytime Functioning Scale

DETAILED DESCRIPTION:
The hypothesis of this investigation is that the BiPAP® Auto with Bi-Flex® improves acceptance of and adherence to positive pressure therapy in participants who are newly diagnosed with OSA and who meet objective criteria for PAP failure during their initial encounter with CPAP in the sleep laboratory.

This hypothesis will be tested using a two-arm, randomized, double-blind design. Participants failing to tolerate CPAP therapy in the sleep laboratory during their titration night will be randomized to a BiPAP® Auto with Bi-Flex® titration or a CPAP titration night in the lab. Participants will then go home with their respective therapy for three months.

ELIGIBILITY:
Inclusion Criterion:

1. Age 21-75
2. New Diagnosis of OSA with a baseline RDI ≥ 15 events/hr of sleep determined by either full night or split night PSG
3. Able and willing to provide written informed consent
4. Able to follow study procedures
5. Sub-optimal PSG titration with at least 3 hours of attempted PAP titration (defined below): and deemed by their physician as a titration failure

Sub-optimal PSG titration: at least one of the following:

1. Poor sleep efficiency during titration period (sleep efficiency ≤ 70%) (participants may be on sleep medications as per standard lab CPAP protocol ) or;
2. Frequent arousals based on three seconds of alpha frequency on EEG (non PLM-related) of 20 or greater per hour during the titration portion of the study or;
3. CPAP titration aborted due to participant's request (due to intolerance), or
4. Persistent sleep disruption despite therapeutic CPAP therapy and in the judgment of the reviewing physician, suggesting a low probability to CPAP adherence

Exclusion Criterion:

1. Participation in another interventional research study within the last 30 days
2. Major uncontrolled medical or psychiatric condition such as congestive heart failure, neuromuscular disease, renal failure etc.
3. Prior CPAP or Bi-Level PAP use (within last 2 years)
4. Chronic respiratory failure or insufficiency, moderate COPD (FEV1 < 60%), or any known condition of an elevation of arterial carbon dioxide levels while awake
5. Surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days
6. Presence of an untreated, diagnosable, non-OSA related sleep disorder (e.g. restless legs syndrome, insomnia, etc.)
7. Periodic Limb movement arousal index of 10 or greater.
8. Refusal to consider further interventions to standard CPAP to optimize positive pressure therapy (e.g. different mask than what was used in lab)
9. PAP therapy otherwise medically complicated or contraindicated such as those with a difficult to size or adjust interface (mask) resulting in facial pain, skin irritation or trauma, or excessive air leaks
10. Shift workers or people experiencing jet lag
11. Known history of alcohol and or drug abuse
12. Diagnosis of Complex Sleep Apnea, (appears to be classic obstructive or mixed sleep apnea, but exhibits disruptive central apneas and periodic breathing on CPAP) 11, 12 or persistent central apnea during diagnostic PSG.
13. Diagnosis of Attention Deficit Hyperactivity Disorder
14. Chronic Hypnotic use (nightly use for three months or less)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
proportion of participants compliant (at least four hours of use per night for all nights) in the Auto Bilevel group compared to the CPAP group after 90 days of treatment during the investigation. | 90 days

SECONDARY OUTCOMES:
ASdherence to BiPAP® Auto with Bi-Flex® therapy compared to CPAP therapy will include: compliance, AHI, HRV, FOSQ, Visual Analog Scale for mask comfort & satisfaction, ESS, PVT, Attitudes toward use, Actigraphy & sleep diary, FSS, & DFS | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Clayton Slep Institute, St Louis, Missouri, United States

REFERENCES:
- [Derived] Powell ED, Gay PC, Ojile JM, Litinski M, Malhotra A. A pilot study assessing adherence to auto-bilevel following a poor initial encounter with CPAP. J Clin Sleep Med. 2012 Feb 15;8(1):43-7. doi: 10.5664/jcsm.1658. PMID 22334808